CLINICAL TRIAL: NCT03354026
Title: Clinical Evaluation of Removing Blood Stasis Therapy in Treating Acute Cerebral Hemorrhage Safety and Efficacy
Acronym: CERBSTTSCH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Collaborators: Lianjiang people's Hospital (Unknown); Shenyang Second Hospital of traditional Chinese Medicine (Unknown); The Third People's Hospital of Hubei Province (Other); Liaocheng People's Hospital (Other); Zengcheng Hospital of traditional Chinese Medicine (Unknown); Shouguang people's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JDZX2015048
Record Dates: First submitted 2017-11-10; First posted 2017-11-27 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Intracerebral Hemorrhage, Hypertensive; Traditional Chinese Medicine
Keywords: Blood-breaking Decotion
MeSH Terms: conditions — Intracranial Hemorrhage, Hypertensive | interventions — Phytotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Our randomized program was completed by the key research laboratory of clinical research from the Traditional Chinese medicine Hospital of Guangdong Province. We design 306 cases into three groups: Group A, B, C in the proportion of 1:1:1. Group A is the experimental group used RBS, which include 8 herbals. Group B is the experimental group used PBS, which include all the herbals in Group A except Leech and Tabanus, rhubarb. Group C is a placebo group. This study adopts a stratified random sampling method and intra slice randomization on the basis of using PROC PLAN progress on SAS V9.2. On the other hand, this trial measures and the control measures will be made blind doubly. The surface of the opaque random envelopes will indicate the information of the test name, hospital name and the entry sequence number of patient. The research process of incorporating patient, dispensing medicine depending on the random envelopes and ect will all be supervised by the researchers each other.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: AICH-PXZY (Experimental): Removing Blood Stasis medicine with folium sennae , Polygonum cuspidatum and so on, 8 herbals, Tong-fu-xing-shen. The intervention in this group includes po AICH-PXZY bid and the routine treatment of Western Medicine.Torn the medicine bag and take it after mixing with 50-80ml warm water（Or take by nasal feeding).
  Interventions: Drug: AICH-PXZY; Drug: AICH-without PXZY; Drug: AICH-placebo
- Experimental: AICH-without PXZY (Experimental): Removing Blood Stasis medicine without folium sennae and Snakegourd seed, 6 herbals, without the effect of Poxuezhuyu. The intervention in this group includes po AICH-without PXZY bid and the routine treatment of Western Medicine.Torn the medicine bag and take it after mixing with 50-80ml warm water（Or take by nasal feeding).
  Interventions: Drug: AICH-PXZY; Drug: AICH-without PXZY; Drug: AICH-placebo
- Placebo: AICH-placebo (Placebo Comparator): The placebo is made up of Starch, bitter taste and cyclodextrin. The intervention in this group includes po AICH-placebo bid and the routine treatment of Western Medicine.Torn the medicine bag and take it after mixing with 50-80ml warm water（Or take by nasal feeding).
  Interventions: Drug: AICH-PXZY; Drug: AICH-without PXZY; Drug: AICH-placebo

INTERVENTIONS:
Drug: AICH-PXZY — 8herbals (with 2 herbals of Activating blood stagnation and expelling blood stasis herbs) one dose, bid, for 10 days
  Other Names: herbal medicine with Hirudo, Tabanus
Drug: AICH-without PXZY — AICH-2(herbal medicine without Hirudo, Tabanus) (6herbals, without 2 herbals of promoting blood stasis) one dose, bid, for 10 days
  Other Names: herbal medicine without Hirudo, Tabanus
Drug: AICH-placebo — The placebo is made up of Starch, bitter taste and cyclodextrin
  Other Names: Placebo

SUMMARY:
The purpose of this research is to use the "Removing Blood Stasis Decotion" of traditional Chinese medicine treating the acute stage of cerebral hemorrhage with stroke associated pneumonia to explore the impact of "Removing Blood Stasis Therapy" on intestinal microbial flora either within the time window from 6 to 72 hours onset.

DETAILED DESCRIPTION:
objective: to investigate the impact and immunologic mechanism of using the "Removing Blood Stasis Decotion" treatment in SAP after Acute Cerebral Hemorrhage with the concept of Intestinal Micro Ecological Regulation.

Methods: from 2017.01 to 2022.12, 240 cases of AICH, 306 cases of hypertension will be included in 7 research centers. The AICH patients are randomly into 3 groups within 6 to 72hrs from onset, thus there are 3 groups and the treatment will last for 10 days: group A，Removing Blood Stasis herbal medicine(8 herbals); Group B, herbal medicine without Poxuezhuyu activating herbal(6 herbals); Group C, placebo medicine of Chinese medicine.All the patients will be treated according AHA guideline of AICH and will be set to the brain CT and chest X-ray at the onset, 24h later and 10-14days after treatment. The venous blood，feces Specimen and the sputum will be collected in the time point of 6 to 72hrs within onset , 24h later, and 10-14days after treatment.So the rate of enlargement of brain hematoma and the development of SAP in the 72h later, mortality rate in the two weeks and the disability rate in the 90 days can be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years old while younger than 80 years old
* acute cerebral hemorrhage confirmed by brain CT scan within 6 to72 hours from onset
* GCS≥6
* Sign the informed consent form

Exclusion Criteria:

* Tests have confirmed that cerebral hemorrhage caused by brain tumor, blood diseases, cerebrovascular malformation (anomaly) or aneurysm, etc;
* patients with Severe heart, liver and renal insufficiency.
* Intolerance to traditional Chinese medicine (TCM), allergic constitution.
* patients with severe cerebral hernia in the early onset
* Compliance is poor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Hematoma enlargement | 6-72h within onset, 24hrs, 10-14days
  The hematoma volume enlarged 33% or increased 12.5ml defined as hematoma enlargement which are compared with the two CT scans(6-72h within onset and 24h after onset,or 6-72h within onset and 10-14days)

SECONDARY OUTCOMES:
GCS scoring scale | 6-72hours within onset, 24hours later, 3 months
  The Glasgow score was used to assess the coma index.
National Institute of Health of stroke scale | 6-72hours within onset, 24hours later, 3 months
  The NIHSS is for evaluation of neurological deficits.
BI index | 3 months
  BI index <90 defines life cannot be independent. The percentage of BI 100-90 points in the three groups was statistically followed up by 90ds.
Social function activity questionnaire(FAQ) | 3 months
  FAQ is mainly to know the quality of life and living habits of the patients and their families.
fatality rate | 3 months
  Any cause of death within the entire treatment 10ds and follow-up 90ds.
modified rankin scale | 3 months
  Scoring 2-5 is defined as disability, which can be divided into 4 grades: mild, moderate, severe and severe. The percentage of mRS 0-1 points in the three groups will be statistically followed up by 90ds.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Guangdong Provincial Science and Technology Agency, Guangzhou, Guangdong
  - Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided
We will keep the IPD in secret and share that only when the agreement are shown by the Ethics committee and the project committee，including the examination results, genotype, etc.

REFERENCES:
- [Derived] Zhang Q, Zeng L, Chen X, Zhou Y, Gong B, Li H, Guo J. Clinical Evaluation of Herbal Medicine (ICH-012) in Treating Acute Cerebral Haemorrhage: Safety and Efficacy from 6- to 72-Hour Time Window (CRRICHTrial-II). Evid Based Complement Alternat Med. 2018 Aug 26;2018:3120179. doi: 10.1155/2018/3120179. eCollection 2018. PMID 30224926